CLINICAL TRIAL: NCT05393713
Title: Phase 1 Study of the Administration of STI-3031 (Anti-PDL1) Intra-Lymphatically Using the Sofusa® DoseConnect™ DEVICE in Patients With In-Transit Melanoma (Sofusa-2)
Brief Title: Intra-Lymphatic STI-3031 Using the Sofusa DoseConnect Device for Treatment of In-Transit Melanoma, The Sofusa-2 Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low/slow accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC210705; NCI-2022-03440 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-010150 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-05-19; First posted 2022-05-26 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Clinical Stage III Cutaneous Melanoma AJCC v8; Melanoma; Metastatic Melanoma; Recurrent Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — IMC-001; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (STI-3031) (Experimental): Patients receive STI-3031 intra-lymphatically via the DoseConnect device over 1-8 hours QW on days 1, 8, 15, 22, 29, and 36 of cycle 1, and Q2W on days 1, 15, and 29 of cycle 2. Treatment repeats every 42 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR at the end of cycle 2 receive 1-2 additional cycles in the absence of disease progression or unacceptable toxicity. Patients with PR or SD at the end of cycle 2 continue treatment for a total of 9 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anti-PD-L1 Monoclonal Antibody IMC-001; Procedure: Punch Biopsy

INTERVENTIONS:
Biological: Anti-PD-L1 Monoclonal Antibody IMC-001 — Given intra-lymphatically via DoseConnect device
  Other Names: IMC 001; IMC-001; IMC001; STI 3031; STI-3031; STI3031
Procedure: Punch Biopsy — Undergo punch biopsy
  Other Names: BIOPSY, PUNCH; Punch Biopsy of Skin

SUMMARY:
This phase Ib trial tests the safety, side effects, and best dose of STI-3031 given directly into the into the lymph nodes or the lymph vessels (intra-lymphatic) using the Sofusa DoseConnect device in treating patients with melanoma that has spread through a lymph vessel and begins to grow more than 2 centimeters away from the primary tumor but before it reaches the nearest lymph node (in-transit). Immunotherapy with monoclonal antibodies, such as STI-3031, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility, safety, and maximum tolerated dose (MTD) of anti-PD-L1 monoclonal antibody IMC-001 (STI-3031) that can be administered through the DoseConnect device in patients with metastatic melanoma demonstrating in-transit and/or regional lymph node metastases.

SECONDARY OBJECTIVE:

I. To assess clinical benefit rates to STI-3031 administered via DoseConnect device in patients with melanoma in-transit and/or reginal lymph node metastases.

CORRELATIVE OBJECTIVES:

I. To assess lymphatic drainage of the affected extremity via intralymphatic indocyanine green (ICG) prior to first treatment cycle and prior to last treatment cycle.

II. To assess for changes in antitumor immunity as a result of therapy.

OUTLINE:

Patients receive STI-3031 intra-lymphatically via the DoseConnect device over 1-8 hours once weekly (QW) on days 1, 8, 15, 22, 29, and 36 of cycle 1, and once every 2 weeks (Q2W) on days 1, 15, and 29 of cycle 2. Treatment repeats every 42 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients with complete response (CR) at the end of cycle 2 receive 1-2 additional cycles in the absence of disease progression or unacceptable toxicity. Patients with partial response (PR) or stable disease (SD) at the end of cycle 2 continue treatment for a total of 9 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 2-4 weeks, 90 days and every 3 months for up to 2 years after study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Disease characteristics:

  * Newly diagnosed, recurrent, or previously treated in-transit metastatic melanoma (ITM) confined to a single limb with or without regional lymph node involvement

    * For patients with ITM, one of the following must be true:

      * A visible superficial ITM, non-nodal lesion with longest diameter >= 1.0 cm in diameter as assessed using a ruler (e.g., skin nodules) NOTE: Documentation by color photography, including a ruler is required OR
      * A malignant regional lymph node with short axis > 1.0 cm as assessed by computed tomography (CT) scan (CT scan slice thickness recommended to be no greater than 5 mm) OR
      * A non-visible, non-nodal soft tissue mass of the involved extremity with longest diameter >= 1.0 cm as measured with CT scan, CT component of a positron emission tomography (PET)/CT, or magnetic resonance imaging (MRI)
  * Newly diagnosed, recurrent or previously treated metastatic melanoma of the lymph nodes in lymphatic beds accessible to limb-lymphatic infusion (Example: lower limb lymphatic accessible femoral, inguinal pelvic and/or retroperitoneal lymph node metastases; upper limb: axillary, infraclavicular and/or subclavian lymph node metastases)

    * For patients with lymph node metastases only (non ITM) the following must be true:

      * At least one tumor involved lymph nodes must be >= 15 mm as assessed by CT, PET or MRI (target lesion by Response Evaluation Criteria in Solid Tumors [RECIST])
* Hemoglobin >= 8.0 g/dL (obtained =< 15 days prior to registration)
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 15 days prior to registration)
* Platelet count >= 75,000/mm^3 (obtained =< 15 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 15 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 3.0 x ULN (obtained =< 15 days prior to registration)
* Serum creatinine =< 2.0 × ULN (obtained =< 15 days prior to registration)
* Calculated creatinine clearance >= 40 ml/min using the Cockcroft-Gault formula (obtained =< 15 days prior to registration)
* Prothrombin time (PT)/international normalized ratio (INR)/partial thromboplastin time (PTT, aPTT) PT/INR/aPTT =< 1.5 × ULN or if patient is receiving anticoagulant therapy INR or aPTT is within target range of therapy (Within 15 days prior to registration)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only.
* Persons able to become pregnant or able to father a child must be willing to use an adequate method of contraception while on treatment and for 180 days (6 months) after last treatment dose on this study
* Provide written informed consent
* Rochester only: Willingness to provide mandatory blood specimens for correlative research
* Willingness to provide mandatory tissue specimens for correlative research
* Willing to return to enrolling institution for 3-month follow-up (during the Active Monitoring Phase of the study)

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic, and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
  * Persons expecting to conceive or father children during the study or within 180 days (6 months) after the last treatment on this study
* Metastatic melanoma beyond in-transit metastases (ITM) and regional lymph nodes (LNs) that cannot be accessed by intralymphatic infusion by DoseConnect (example: visceral or active central nervous system [CNS] metastatic disease)
* ITM involving the hands and feet (not accessible to DoseConnect infusion)
* ITM NOT involving a limb (i.e., head, neck, or trunk)
* Prior radiation of ITM that are being evaluated as measurable lesions
* Any of the following prior therapies:

  * Allogeneic hematopoietic stem cell transplantation (HSCT)
  * Solid organ transplantation
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy.

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Active autoimmune disease requiring systemic treatment < 2 years prior to registration, documented history of severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents with use of disease modifying agents, corticosteroids, or immunosuppressive drugs

NOTE: Exceptions are allowed for the following conditions:

* Vitiligo
* Resolved childhood asthma/atopy
* Intermittent use of bronchodilators or inhaled steroids
* Daily steroids at dose of =< 10mg of prednisone (or equivalent)
* Local steroid injections
* Stable hypothyroidism on replacement therapy
* Stable diabetes mellitus on therapy (with or without insulin)
* Sjogren's syndrome
* Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) which is not considered a form of systemic treatment and is allowed

  * Uncontrolled intercurrent illness including, but not limited to:
* Ongoing or active infection requiring systemic therapy
* Interstitial lung disease
* Serious, chronic gastrointestinal conditions associated with diarrhea (e.g., Crohn's disease or others)
* Known history of hepatitis B (i.e., known positive hepatitis B virus [HBV] surface antigen [HBsAg] reactive)
* Known active hepatitis C (i.e., positive for hepatitis C virus [HCV] ribonucleic acid [RNA] detected by polymerase chain reaction [PCR])
* Known active tuberculosis (TB)
* Symptomatic congestive heart failure
* Unstable angina pectoris
* Unstable cardiac arrhythmia or
* Psychiatric illness/social situations that would limit compliance with study requirements (e.g., known substance abuse)

  * Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
  * History of severe hypersensitivity reactions to other monoclonal antibodies or known hypersensitivity to the study intervention or its excipients, indocyanine green (ICG) dye or iodine
  * Prior history of Grade 4 immune related adverse event (irAE) with prior immune checkpoint inhibitor (ICI) therapy or failure to recover (< Grade 1) from immune-related adverse event(s) from prior ICI therapy
  * Failure to recover from any adverse events related to any of the following therapies received prior to registration:
* Chemotherapy
* Immunotherapy
* Targeted therapies (e.g., dabrafenib)
* Other investigational agents
* Radiation therapy
* Minor surgical or interventional procedure (NOTE: Biopsy of same limb for diagnosis is allowed)
* Major surgical procedure

  * Previously untreated metastatic melanoma (visceral or CNS). NOTE: Patients with previously treated systemic and CNS melanoma who have been free of disease at systemic sites for >= 12 weeks are eligible for treatment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-02-16 (Actual); Study Completion 2025-02-16 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of STI-3031 that can be administered through the DoseConnect device | Up to 42 days (Cycle 1)
  MTD is the dose level where at most 1 of the 6 patients treated at that dose level develops a dose limiting event (DLE) during the first cycle of treatment and neither a Grade 3 or worse AE attributable to either drug or device or a Grade 2 or worse adverse event (AE) lasting >= 1 week and attributable to device is reported after the first cycle of treatment.
Incidence of adverse events | Up to 2 years
  The maximum grade of each type of adverse event will be recorded for each patient. For each adverse event reported by dose level, the percentage of patients developing any degree of that adverse event as well as the percentage of patients developing a severe degree (Grade 3 or higher) will be determined.

SECONDARY OUTCOMES:
Clinical benefit rate | Up to the end of cycle 3 (126 days)
  Defined as the number of patients who complete 3 cycles of treatment and whose objective tumor status by Response Evaluation Criteria in Solid Tumors (RECIST) is stable, partial response (PR) or complete response (CR) post discontinuation among all eligible patients enrolled.
Progression-free survival (PFS) | From study entry to the documentation of disease progression, assessed up to 2 years
  If a patient dies without a recurrence documented, the patient will be censored at the date of their last disease evaluation unless there is documentation that the patient was progression-free within 3 months of death. PFS distribution will be estimated using the Kaplan-Meier method.
Response rate | Up to 2 years
  Defined as the proportion of patients whose tumor meets the criteria for PR or CR on two consecutive evaluations at least 12 weeks apart among all eligible patients who began treatment.

OTHER OUTCOMES:
Lymphatic flow rate | Baseline and prior to cycle 3
  Descriptive analysis will be performed to report these findings.
Indocyanine green (ICG) lymphography classification | Up to 2 years
  The ICG lymphography classification of the functional status of the lymphatic system first described by Yamamoto et al (Yamamoto 2011) will be utilized. Utilizing descriptive statistics, we will note any changes in the ICG flow patterns and if any improvement or deterioration appears associated with in-transit metastasis (ITM) response, stability, or progressive disease. This work will be exploratory and hypothesis generating.

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios Dimou, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials